CLINICAL TRIAL: NCT01145560
Title: A MultiCentre, Randomized, Double-blind, Placebo-controlled Phase IIb Study to Compare the Efficacy and Safety of Two Dosing Regimens of Intravenous Infusions of AZD9773 (CytoFab™) in Adult Patients With Severe Sepsis and/or Septic Shock
Brief Title: A Study to Compare the Efficacy and Safety of 2 Dosing Regimens of IV Infusions of AZD9773 (CytoFab™) With Placebo in Adult Patients With Severe Sepsis and/or Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D0620C00003
Record Dates: First submitted 2010-06-07; First posted 2010-06-16 (Estimated); Results first posted 2013-09-23 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-09

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: severe sepsis; TNF neutralisation; septic shock patients
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — AZD9773; CytoFab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- 1 (Experimental): AZD9773 250/50 units/kg
  Interventions: Drug: AZD9773
- 2 (Experimental): AZD9773 500/100 units/kg
  Interventions: Drug: AZD9773
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9773 — A single loading dose following by up to 9 maintenance doses; doses to be given every 12 hours over a period of 5 days
  Other Names: CytoFab™
  Arms: 1; 2
Drug: Placebo — Placebo
  Arms: 3

SUMMARY:
The primary purpose of this study to evaluate the effect of two different doses of AZD9773 (CytoFab™) versus placebo on ventilator free days (VFDs) over the first 28 days after the start of dosing with AZD9773 in patients with severe sepsis and/or septic shock, who are already receiving appropriate standard of care treatment for sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a first episode of sepsis during this hospitalisation and objective evidence of infection that requires parenteral antibiotics.
* At least 2 of 4 SIRS criteria in the 24 hours before organ dysfunction (must include either fever OR elevated white blood cells [WBC])
* Cardiovascular or respiratory dysfunction.

Exclusion Criteria:

* Immunocompromising comorbidities or concomitant medications:

  1. Advanced human immunodeficiency virus (HIV) infection (CD4 ≤50/mm3).
  2. Stage III or IV cancer.
  3. Haemopoietic or lymphoreticular malignancies not in remission.
  4. Receiving radiation therapy or chemotherapy.
  5. Stem cell, organ or bone marrow transplant in the past 6 months.
  6. Absolute neutrophil count <500 per μL.
  7. High dose steroids or other immunocompromising drugs.
* Concomitant diseases:

  1. Deep seated fungal infection or active tuberculosis.
  2. Cirrhosis with portal hypertension or Childs-Pugh Class C.
  3. History of chronic hypercarbia, respiratory failure in past 6 months or use of home oxygen in the setting of severe chronic respiratory disease.
  4. Neuromuscular disorders that impact breathing/spontaneous ventilation.
  5. Quadriplegia.
  6. Cardiac arrest in the past 30 days.
  7. New York Heart Association functional Class IV due to heart failure or any disorder.
  8. Burns over > 30% of body surface area.
* Medication and allergy disqualifications.

  1. Treatment with anti-TNF agents within the last 8 weeks.
  2. Previously received ovine derived products (CroFab™, DigiFab™).
  3. Sheep product allergy or allergy to latex, papain, chymopapain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Bernard, MD, Principal Investigator — Vanderbilt University; Warren Botnick, MD, Study Director — Parexel; Justin Lindemann, MD, Study Director — AstraZeneca; Wayne Dankner, MD, Study Director — Parexel; Jiri Juchelka, MD, Study Director — Parexel
Locations (52):
- Australia (9):
  - Research Site, Blacktown, New South Wales
  - Research Site, Wollongong, New South Wales
  - Research Site, Herston, Queensland
  - Research Site, Nambour, Queensland
  - Research Site, Woollongabba, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Clayton, Victoria
  - Research Site, Footscray, Victoria
  - Research Site, Fremantle, Western Australia
- Belgium (6):
  - Research Site, Antwerp, Belgium
  - Research Site, Brussels, Belgium
  - Research Site, Genk, Belgium
  - Research Site, Godinne, Belgium
  - Research Site, Liège, Belgium
  - Research Site, Ottignies, Belgium
- Canada (8):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Halifax, Nova Scotia
  - Research Site, Ottawa, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Québec, Quebec
- Czechia (3):
  - Research Site, Hradec Králové
  - Research Site, Prague
  - Research Site, Ústí nad Labem
- Finland (2):
  - Research Site, Kuopio
  - Research Site, Tampere
- France (15):
  - Research Site, Angers
  - Research Site, Dijon
  - Research Site, La Roche-sur-Yon
  - Research Site, Limoges
  - Research Site, Montauban
  - Research Site, Nantes
  - Research Site, Nîmes
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Saint-Michel
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Vandœuvre-lès-Nancy
- Spain (9):
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Sabadell, Barcelona
  - Research Site, Barcelona, Catalonia
  - Research Site, Terrassa, Catalonia
  - Research Site, Santiago de Compostela, Coruna
  - Research Site, Getafe, Madrid
  - Research Site, Madrid, Madrid
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Valencia, Valencia

REFERENCES:
- [Derived] Yates JW, Das S, Mainwaring G, Kemp J. Population pharmacokinetic/pharmacodynamic modelling of the anti-TNF-alpha polyclonal fragment antibody AZD9773 in patients with severe sepsis. J Pharmacokinet Pharmacodyn. 2012 Dec;39(6):591-9. doi: 10.1007/s10928-012-9270-4. Epub 2012 Sep 23. PMID 23001587
- See also: CSR-D0620C00003.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1665&filename=CSR-D0620C00003.pdf
- See also: redacted-CSP-D0620C00003.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1665&filename=Global_Ph_2b-D0620C00003_redated_text_18_July_2014.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled from approximately 100 centres worldwide.
Groups:
- AZD9773 250/50 Units/kg: AZD9773 250/50 units/kg IV
- AZD9773 500/100 Units/kg: AZD9773 500/100 units/kg IV
- Placebo: Saline
Period: Overall Study
Arm/Group | AZD9773 250/50 Units/kg | AZD9773 500/100 Units/kg | Placebo
Started | 100 | 100 | 100
Received Treatment | 99 | 98 | 99
Completed Treatment | 69 (9 patients died during the treatment period without completing the full course of treatment.) | 85 (8 patients died during the treatment period without completing the full course of treatment.) | 78 (7 patients died during the treatment period without completing the full course of treatment.)
Completed | 96 (20 patients died during the study. Death was not a reason for treatment or study discontinuation.) | 96 (33 patients died during the study. Death was not a reason for treatment or study discontinuation.) | 98 (27 patients died during the study. Death was not a reason for treatment or study discontinuation.)
Not Completed | 4 | 4 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — No study drug by 24h after organ failure | 1 | 0 | 0
Not completed — Accidental unblinding of study treatment | 0 | 1 | 0
Not completed — False insurance information | 0 | 1 | 0
Not completed — Withdrawal of therapy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD9773 250/50 Units/kg | AZD9773 500/100 Units/kg | Placebo | Total
Number analyzed (Participants) | 100 | 100 | 100 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (15.76) | 66.6 (14.61) | 64.1 (15.25) | 65.0 (15.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 32 | 112
  Male | 60 | 60 | 68 | 188

OUTCOME MEASURES:

1. Primary Outcome: Ventilator-free Days (VFDs) Over 28 Days
Description: Number of ventilator-free days (VFDs)
Time Frame: Over 28 days following first dose
Population: Intention-to-treat analysis set
Measure: Median (Full Range); unit: Days
Arm/Group | AZD9773 250/50 Units/kg | AZD9773 500/100 Units/kg | Placebo
Number analyzed (Participants) | 100 | 100 | 100
Days | 21.0 [0 to 28] | 17.5 [0 to 28] | 19.0 [0 to 28]

2. Secondary Outcome: 7-day Mortality
Description: Number of patients who died over 7 days
Time Frame: Over 7 days following first dose
Population: Intention-to-treat analysis set
Measure: Number; unit: Participants
Arm/Group | AZD9773 250/50 Units/kg | AZD9773 500/100 Units/kg | Placebo
Number analyzed (Participants) | 100 | 100 | 100
Participants | 9 | 9 | 10

3. Secondary Outcome: 28-day Mortality
Description: Number of patients who died over 28 days
Time Frame: Over 28 days following first dose
Population: Intention-to-treat analysis set
Measure: Number; unit: Participants
Arm/Group | AZD9773 250/50 Units/kg | AZD9773 500/100 Units/kg | Placebo
Number analyzed (Participants) | 100 | 100 | 100
Participants | 15 | 27 | 20

4. Secondary Outcome: Safety and Tolerability
Description: Number of patients with treatment-emergent adverse events
Time Frame: All study visits (over 90 days following first dose)
Population: Safety Analysis Set
Measure: Number; unit: Participants
Arm/Group | AZD9773 250/50 Units/kg | AZD9773 500/100 Units/kg | Placebo
Number analyzed (Participants) | 100 | 97 | 99
Participants | 86 | 87 | 92

ADVERSE EVENTS:
Description: One patient received incorrect dose of AZD9773, which explains the difference between the 2 AZD9773 dose groups for the patients in the following tables for adverse events.
Arm/Group | AZD9773 250/50 Units/kg | AZD9773 500/100 Units/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 28/100 | 27/97 | 31/99
Other Adverse Events (participants affected / at risk) | 74/100 | 71/97 | 68/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD9773 250/50 Units/kg (N=100) | AZD9773 500/100 Units/kg (N=97) | Placebo (N=99)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 2
Cardiac Arrest (Cardiac disorders) | 0 | 1 | 1
Cardiac Failure Acute (Cardiac disorders) | 0 | 1 | 0
Cardiogenic Shock (Cardiac disorders) | 0 | 1 | 0
Sick Sinus Syndrome (Cardiac disorders) | 0 | 1 | 0
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Fistula (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 2 | 1
Gastrointestinal Necrosis (Gastrointestinal disorders) | 1 | 1 | 0
Intestinal Infarction (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 0 | 1 | 2
Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatic Fistula (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Multi-Organ Failure (General disorders) | 0 | 3 | 3
Pyrexia (General disorders) | 0 | 0 | 1
Biliary Tract Disorder (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cytolytic Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic Lesion (Hepatobiliary disorders) | 0 | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Abdominal Wall Abscess (Gastrointestinal disorders) | 0 | 0 | 1
Aspergillosis (Infections and infestations) | 0 | 0 | 1
Device Related Sepsis (Infections and infestations) | 1 | 0 | 1
Empyema (Infections and infestations) | 1 | 0 | 0
Encephalitis Herpes (Infections and infestations) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Fungal Oesophagitis (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Infectious Peritonitis (Infections and infestations) | 0 | 1 | 1
Meningitis Staphylococcal (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 5
Sepsis (Infections and infestations) | 2 | 1 | 1
Septic Shock (Infections and infestations) | 2 | 2 | 1
Systemic Candida (Infections and infestations) | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0
Splenic Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Autonomic Nervous System Imbalance (Nervous system disorders) | 0 | 1 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Critical Illness Polyneuropathy (Nervous system disorders) | 0 | 0 | 1
Guillain-Barre Syndrome (Nervous system disorders) | 1 | 0 | 0
Hepatic Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0
Abnormal Behaviour (Psychiatric disorders) | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1
Respiratory Gas Exchange Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash Vesicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Air Embolism (Vascular disorders) | 1 | 0 | 0
Extremity Necrosis (Vascular disorders) | 0 | 1 | 1
Ischaemia (Vascular disorders) | 0 | 0 | 1
Shock (Vascular disorders) | 2 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD9773 250/50 Units/kg (N=100) | AZD9773 500/100 Units/kg (N=97) | Placebo (N=99)
Anaemia (Blood and lymphatic system disorders) | 20 | 18 | 22
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 4 | 4
Atrial Fibrillation (Cardiac disorders) | 11 | 14 | 8
Constipation (Gastrointestinal disorders) | 7 | 11 | 9
Diarrhoea (Gastrointestinal disorders) | 12 | 9 | 14
Nausea (Gastrointestinal disorders) | 5 | 2 | 7
Vomiting (Gastrointestinal disorders) | 5 | 2 | 5
Generalised Oedema (General disorders) | 6 | 2 | 4
Oedema (General disorders) | 4 | 2 | 5
Oedema Peripheral (General disorders) | 3 | 3 | 5
Pyrexia (General disorders) | 6 | 5 | 5
Pneumonia (Infections and infestations) | 5 | 4 | 7
Urinary Tract Infection (Infections and infestations) | 2 | 6 | 7
Fluid Overload (Metabolism and nutrition disorders) | 3 | 5 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 3 | 5
Hypernatraemia (Metabolism and nutrition disorders) | 6 | 3 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 1 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 9 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 2 | 6
Agitation (Psychiatric disorders) | 6 | 7 | 8
Anxiety (Psychiatric disorders) | 6 | 1 | 7
Confusional State (Psychiatric disorders) | 7 | 4 | 5
Insomnia (Psychiatric disorders) | 5 | 3 | 11
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 4
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 4 | 5 | 6
Rash (Skin and subcutaneous tissue disorders) | 5 | 3 | 4
Hypertension (Vascular disorders) | 5 | 5 | 7
Hypotension (Vascular disorders) | 4 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less